CLINICAL TRIAL: NCT04003090
Title: Evaluation of Citicoline Concentration in Human Vitreous After Topical Administration: a Cross-sectional Study
Brief Title: Citicoline Concentration in Human Vitreous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto di Ricerca Neuroftalmologia S.r.l. (Network)
Collaborators: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N.61/17/FB
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2018-03

CONDITIONS: Neurodegenerative Diseases
Keywords: ophthalmic solution; glaucoma; retinal ganglion cells; neuroprotective effect
MeSH Terms: conditions — Neurodegenerative Diseases; Glaucoma | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Citicoline eyes (Experimental): Patients had to administer 3 drops/day of an ophthalmic solution containing citicoline 1% eye-drops, 0.2% high molecular weight hyaluronic acid and 0.01% benzalkonium chloride for 14 days before surgery and 2 hours prior to surgery.
  Interventions: Drug: Citicoline

INTERVENTIONS:
Drug: Citicoline — After treatment with a solution containing citicoline 1% eye-drops, 0.2% high molecular weight hyaluronic acid and 0.01% benzalkonium chloride patients underwent a 23G standard 3-port pars plana vitrectomy. The vitreous sample was taken at the beginning of the surgery and then analyzed.

SUMMARY:
Elegible patients were included in the study and underwent treatment with a solution of citicoline 1% eye-drops, 0.2% high molecular weight hyaluronic acid and 0.01% benzalkonium chloride prior to surgery. The vitreous samples were taken at the beginning of the surgery and analyzed for qualitative/quantitative determination of vitreous concentration of citicoline and its metabolites by means of high performance liquid chromatography.

DETAILED DESCRIPTION:
At the visit all patients underwent comprehensive ophthalmological examination including best corrected visual acuity assessment, slit lamp evaluation, IOP measurement using Goldmann applanation tonometry, and fundus dilated indirect ophthalmoscopy.

Additionally, all patients had central retinal thickness measurements with spectral-domain optical coherence tomography associated with central corneal thickness (CCT) and corneal endothelial cells density (ECD) evaluations.

Patients started the treatment with 1 drop of a solution of citicoline 1% eye-drops, 0.2% hyaluronic acid and 0.01% benzalkonium chloride for 3 times/day over a total time of 14 days before surgery and 1 drop 2 hours prior to the surgery.

Five patients served as controls and received a vehicle solution without citicoline.

The primary aim of the study was to evaluate the presence and concentration of citicoline and its metabolites (choline, cytidine and uridine) in the vitreous body in vivo in human eyes after topical eye-drops administration by means of high performance liquid chromatography.

Secondary aims were the comparison of citicoline and its metabolites concentration in the vitreous of treated phakic and pseudophakic eyes and the correlations with age and ocular biometric parameters including CCT and ECD.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ability to understand and sign the written informed consent
* diagnosis of epiretinal membrane (ERM) with surgical indication for pars-plana vitrectomy

Exclusion Criteria:

* laser treatments and ocular surgery in the past 6 months
* hypersensitivity to the active ingredients used in the study
* other systemic or ocular diseases different from ERM that could affect the outcome of the study
* aphakia or previous complicated cataract surgery
* intraocular lens (IOL) in the anterior chamber
* treatment with systemic citicoline or other potential neuroprotective agents in the past 6 months
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Citicoline and metabolites concentration in human vitreous | 14 days
  Evaluate the presence and concentration of citicoline and its metabolites (choline, cytidine and uridine) in the vitreous body in vivo in human eyes after topical eye-drops administration.

SECONDARY OUTCOMES:
Citicoline and metabolites concentration in phakic and pseudophakic eyes | 14 days
  Comparison of citicoline and its metabolites concentration in the vitreous of phakic and pseudophakic eyes and correlations with age, central corneal thickness and corneal endothelial cells density.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Oddone, MD, PHD, Principal Investigator — Fondazione G.B. Bietti, IRCCS
Locations (1):
- Fondazione G.B. Bietti- IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No